CLINICAL TRIAL: NCT02644408
Title: Megestrol Acetate for the Improvement of Quality of Life in Esophageal Cancer With Chemoradiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAIQF
Record Dates: First submitted 2015-11-27; First posted 2015-12-31 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2019-10

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma; Stage II Esophageal Squamous Cell Carcinoma
Keywords: Chemoradiotherapy; Esophageal Squamous Cancer; Megestrol
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy; Radiation; Drug Therapy

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients and the medical professionals who cared for them were unaware of the assigned study regimen.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Megestrol and chemoradiotherapy (Experimental): Megestrol（Yining）：160mg/d，po,5 weeks in total，oen week before chemoradiotherapy and one week after chemoradiotherapy.
  chemoradiotherapy：chemotherapy and radiotherapy： 50Gy in total，2 Gy/d，5d/w.
  Interventions: Drug: Megestrol（Yining）; Radiation: radiotherapy; Other: chemotherapy
- chemoradiotherapy (Active Comparator): chemoradiotherapy：chemotherapy and radiotherapy： 50Gy in total，2 Gy/d，5d/w.
  Interventions: Radiation: radiotherapy; Other: chemotherapy

INTERVENTIONS:
Drug: Megestrol（Yining） — Megestrol（Yining）: 160mg/d, po,7 weeks in total, one week before chemoradiotherapy and one week after chemoradiotherapy.
  Other Names: Yining
  Arms: Megestrol and chemoradiotherapy
Radiation: radiotherapy — radiotherapy (radiation): 50Gy in total，2 Gy/d，5d/w.
  Other Names: radiation
Other: chemotherapy — capecitabine(Aibin)：625mg/m2, bid d1-5; q1w, po,5 weeks in total or capecitabine(Aibin) plus Oxaliplatin(Aiheng)：65mg/m2，d1，8, 22, 29,I.V. or cisplatin: 75mg/m2 d1，29 5-Fu：750mg/m2CIV24h d1-4，d29-32. The 3 regimens were Randomly distributed to patients.

SUMMARY:
Megestrol is a semisynthetic progesterone derivatives, have promote anabolic effects. Can improve appetite, weight gain, and improve bone marrow suppression, increase the tolerance put, chemotherapy, improve the quality of life, is widely used in tumor radiation and chemotherapy of terminally ill patients. But because of its vascular embolization, vaginal bleeding, arrhythmia and other serious complications, there is no unified standard.

The purpose of this study was to evaluate megestrol in esophageal squamous carcinoma radical chemoradiation curative effect and side effects, for rational use in the process of radiation and chemotherapy megestrol provide guidelines. A total of 210 patients will be accrued from China.The primary end point is quality of life (will be evaluated by EORTC QLQ-C30); the secondary end point is the pathological response after treatment and adverse events.

DETAILED DESCRIPTION:
The investigators plan to recruit the patients who were pathologically confirmed with esophageal squamous cell carcinoma and performed chemoradiotherapy from the Oct 2014. The patients will be divided into two groups.Experimental group：esophageal cancer patients with oral megestrol chemoradiation. Megestrol（Yining）：160mg/d，po,5 weeks in total，oen week before chemoradiotherapy and one week after chemoradiotherapy.

chemoradiotherapy：chemotherapy and radiotherapy： 50Gy in total，2 Gy/d，5d/w.Control group: Esophageal cancer patients with chemoradiation without oral megestrol.chemoradiotherapy：chemotherapy and radiotherapy： 50Gy in total，2 Gy/d，5d/w.The primary end point is quality of life (will be evaluated by EORTC QLQ-C30); the secondary end point is the pathological response after treatment and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75years old
* Histologically proven squamous cell carcinoma of the esophagus the tumor was in T2-4N0-2M0
* The patients have not received the surgery or chemo-radiotherapy.
* Hb≥80g/L, absolute neutrophil count ≥1.5×109/L, Plt≥90×109/L,
* ALT、AST≤2.5*N,Cr≤1.5*N.
* performance status score 0-2

Exclusion Criteria:

* Pregnant, lactating women
* Oxaliplatin or fluorouracil Allergy or metabolic disorders
* Radiotherapy contraindications
* History of organ transplantation
* Brain metastasis
* The peripheral nervous system disorders
* Severe infection
* Oral capecitabine who have difficulty with,such as dysphagia,The activities of digestive ulcer, Gastrointestinal bleeding
* Severe chronic diseases, such as, hepatopathy, nephropathy, respiratory disease,high blood pressure, diabetes.
* Other malignant tumor in recent 5 years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoF) | 16 weeks
  evaluated by EORTC QLQ-C30 questionnaire

SECONDARY OUTCOMES:
pathological response | 16 weeks
  complete response(CR)
adverse events | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, MD, PhD, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology; Ruinuo Jia, MD, PhD, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Tanyou Shan, MD, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Xinshuai Wang, MD, PhD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Jiachun Sun, MD, PhD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Guoqiang Kong, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaozhi Yuan, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaoshan Feng, MD, PhD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Zhuo, MD, PhD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Jing Ren, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruina Yang, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Weijiao Yin, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Wei Wang, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yali Zhang, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Wang, MD, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JW, Kim JH, Choi EK, Lee SW, Yoon SM, Song SY, Lee YS, Kim SB, Park SI, Ahn SD. Prognosis of esophageal cancer patients with pathologic complete response after preoperative concurrent chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):691-7. doi: 10.1016/j.ijrobp.2010.06.041. Epub 2010 Oct 1. PMID 20888705
- [Background] Ezeoke CC, Morley JE. Pathophysiology of anorexia in the cancer cachexia syndrome. J Cachexia Sarcopenia Muscle. 2015 Dec;6(4):287-302. doi: 10.1002/jcsm.12059. Epub 2015 Oct 27. PMID 26675762
- [Background] Ordu C, Pilanci KN, Koksal UI, Okutur K, Saglam S, Tecimer C, Demir G. Can megestrol acetate induce thrombosis in advanced oncology patients receiving chemotherapy? Asian Pac J Cancer Prev. 2014;15(23):10165-9. doi: 10.7314/apjcp.2014.15.23.10165. PMID 25556442
- [Background] Kanat O. Management of cancer cachexia (reply). Tumori. 2014 Jan-Feb;100(1):e1. doi: 10.1700/1430.15826. No abstract available. PMID 24675504
- [Background] Greig CA, Johns N, Gray C, MacDonald A, Stephens NA, Skipworth RJ, Fallon M, Wall L, Fox GM, Fearon KC. Phase I/II trial of formoterol fumarate combined with megestrol acetate in cachectic patients with advanced malignancy. Support Care Cancer. 2014 May;22(5):1269-75. doi: 10.1007/s00520-013-2081-3. Epub 2014 Jan 4. PMID 24389826
- [Background] Hong S, Jeong IG, You D, Lee JL, Hong JH, Ahn H, Kim CS. Safety of megestrol acetate in palliating anorexia-cachexia syndrome in patients with castration-resistant prostate cancer. J Korean Med Sci. 2013 May;28(5):687-92. doi: 10.3346/jkms.2013.28.5.687. Epub 2013 May 2. PMID 23678259
- [Background] Argiles JM, Anguera A, Stemmler B. A new look at an old drug for the treatment of cancer cachexia: megestrol acetate. Clin Nutr. 2013 Jun;32(3):319-24. doi: 10.1016/j.clnu.2013.01.004. Epub 2013 Jan 22. PMID 23395103
- [Background] Madeddu C, Dessi M, Panzone F, Serpe R, Antoni G, Cau MC, Montaldo L, Mela Q, Mura M, Astara G, Tanca FM, Maccio A, Mantovani G. Randomized phase III clinical trial of a combined treatment with carnitine + celecoxib +/- megestrol acetate for patients with cancer-related anorexia/cachexia syndrome. Clin Nutr. 2012 Apr;31(2):176-82. doi: 10.1016/j.clnu.2011.10.005. Epub 2011 Nov 1. PMID 22047681
- [Background] Gullett NP, Mazurak VC, Hebbar G, Ziegler TR. Nutritional interventions for cancer-induced cachexia. Curr Probl Cancer. 2011 Mar-Apr;35(2):58-90. doi: 10.1016/j.currproblcancer.2011.01.001. PMID 21420558